CLINICAL TRIAL: NCT01958138
Title: Isoflurane Versus Combination Of Propofol With Isoflurane For Removal Of Laryngeal Mask Airway In Children
Brief Title: Isoflurane Versus Propofol for Removal of LMA in Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dileep Kumar, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1995-Ane-ERC-11
Record Dates: First submitted 2012-06-19; First posted 2013-10-09 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Complication of Anesthesia
Keywords: Laryngeal Mask Airway; Propofol; Isoflurane; Pediatric patients; Emergence
MeSH Terms: interventions — Propofol; Isoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol with Isoflurane (Experimental): Propofol with Isoflurane, Group-I is the intervention arm with combination of two drugs such as low dose propofol and Isoflurane MAC awake.
  Interventions: Drug: comparison of group-I (low dose propofol with isoflurane)
- alone isoflurane (Active Comparator): The group-II is the control arm of study by using the only Isoflurane 1.2 MAC
  Interventions: Drug: comparison of group-I (low dose propofol with isoflurane)

INTERVENTIONS:
Drug: comparison of group-I (low dose propofol with isoflurane) — Prior to LMA removal in group-I, isoflurane MAC awake (MAC less than 0.5) will be achieved in expiratory gases with 60% nitrous oxide and 40% oxygen. Propofol 1 mg/Kg will be combined with Isoflurane MAC awake and LMA will be removed after 20 seconds of propofol administration in group-I. The group-II LMA will be removed at end expiratory isoflurane MAC of 1.2% with 60% nitrous oxide and 40% oxygen
  Other Names: group-II (alone isoflurane MAC 1.2%)

SUMMARY:
The study will be done in paediatric patients by comparing two different techniques of Laryngeal Mask Airway (LMA) removal under deep anesthetic plane.

The both study techniques will be compared for safe LMA removal on the basis of adverse airway events and emergence time duration and recovery room stay timing.

DETAILED DESCRIPTION:
* Study will be start after confirming the approval of institutional ethical review committee and after fulfilling the study inclusion criteria. The detailed study protocol will be explain to the parent/guardian and written & informed consent will be taking on his/her will.
* Inclusion Criteria

  * Age between 2 to 10 years,
  * American Society of Anaesthesiologists (ASA) physical status I & II,
  * Patient is not contraindicated to Laryngeal Mask Airway insertion,
  * Elective below umbilical general surgical procedures
  * patient is planned for general anesthesia with spontaneous breathing.
* Fifty patients will participate in both study groups.
* All patients will be premedicated with oral midazolam 0.3mg/kg, 45 to 60 minutes prior to induction.
* After arrival of patients in operating room, routine anesthesia monitoring will be applied and baseline blood pressure, heart rate, respiratory rate and oxygen saturation will be recorded.
* Patient will be induced with anesthetic induction inhalational agent (sleeping drug) sevoflurane 8% with oxygen by pediatric anesthesia circle system. The sevoflurane concentration will be adjusted to 3% to 4% once the adequate depth of anesthesia achieved, as evident by jaw relaxation and tolerance of an oral airway.
* The LMA will be placed after the insertion of intravenous line.
* The LMA size will be determined as per manufacturer's recommendation; which suggest 1.5 LMA size for 5-10 kg, size 2 for 10-20 kg and size 2.5 for 20-30 kg.
* The anesthesia will be maintained with isoflurane in 60% nitrous oxide and 40% oxygen. Patients will be ventilated by spontaneous mode by 'Mapleson F anesthesia circuit' and for above 25 Kg patient, the circle system will be used.
* Caudal analgesia was standardised in both study groups.
* Prior to LMA removal in group-I, isoflurane MAC awake (MAC less than 0.5) will be achieved in expiratory gases with 60% nitrous oxide and 40% oxygen. Propofol 1 mg/Kg will be combined with Isoflurane MAC awake and LMA will be removed after 20 seconds of propofol administration in group-I.

The group-II LMA will removed at end expiratory isoflurane MAC of 1.2% with 60% nitrous oxide and 40% oxygen. In both groups; LMA will be removed with inflated cuff, throat was suctioned and patients were turned into lateral recovery position.

Isoflurane and nitrous oxide were turned off and 100% oxygen supplemented till the patient had regained consciousness. All participants were transported to Post Anesthesia Care Unit (PACU) once ensured airway patency and peripheral oxygen saturation (Sp02) greater than 93% on room air. Children were allowed to wake up effortlessly in PACU at oxygen 5 litters/minutes via Hudson mask.

- The following study variables will be recorded;

1. Emergence time ( patient awakening time),
2. Duration of recovery room stay (Post anesthesia care unit),
3. Smooth Laryngeal Mask Airway removal will be assessed by

   * Cough,
   * Hypersalivation,
   * 02 desaturation < 90%,
   * Teeth clenching,
   * Airway obstruction requiring jaw support,
   * Laryngospasm,
   * Bronchospasm,
   * Retching,
   * Vomiting,
4. Confounding variables will be assessed like;

   * Patients demographics,
   * Duration of surgery,
   * Duration of anesthesia,
   * Type of surgery,
   * Mode of analgesia
   * Number of Laryngeal Mask Airway insertion attempts:

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist class-I & II patients.
* mallampatis class I & II.
* Age from 2 years to 10 years.
* Elective surgical patients for below umbilical general surgical procedures.

Exclusion Criteria:

* Congenital disorders
* Airway or facial abnormalities
* Reactive airway disease/asthma
* Anticipated difficult airway
* History of Upper respiratory tract infection in last 3 weeks
* History of gastroesophageal reflux disorders
* Known allergic to isoflurane and propofol

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Emergence airway complications | 15 minutes of continuous monitoring and time frame was started from the LMA removal
  Smooth LMA removal will be assessed by adverse airway events like; coughing, bucking, hypersalivation, O2 desaturation (Sp02<90%), airway obstruction (noisy or stridor breathing) requiring jaw support, laryngospasm, bronchospasm, retching and vomiting, time duration from LMA removal up to 15 minutes.
Emergence time duration | 15 minutes of continuous monitoring and time frame was started from the LMA removal
  Impact on emergence time duration because of intervention such as delayed awakening or responding
Post anaesthesia care unit stay time duration | 0-45 minutes of continuous monitoring and time frame was started from the PACU admission to discharge
  Impact of intervention on post anaesthesia care unit admission to discharge time duration

CONTACTS AND LOCATIONS:
Overall Officials: dileep kumar, FCPS, Principal Investigator — Aga Khan University Hospital Karachi
Locations (1):
- Operating room at Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frediani M, Blanchini G, Capanna M, Casini L, Costa M, Uggeri S, Meini M, Pacini P. [The laryngeal mask in pediatric anesthesia]. Minerva Anestesiol. 1996 Mar;62(3):65-71. Italian. PMID 8767151
- [Background] Brain AI. The laryngeal mask--a new concept in airway management. Br J Anaesth. 1983 Aug;55(8):801-5. doi: 10.1093/bja/55.8.801. PMID 6349667
- [Background] Samarkandi AH. Awake removal of the laryngeal mask airway is safe in paediatric patients. Can J Anaesth. 1998 Feb;45(2):150-2. doi: 10.1007/BF03013254. PMID 9512850
- [Background] Splinter WM, Reid CW. Removal of the laryngeal mask airway in children: deep anesthesia versus awake. J Clin Anesth. 1997 Feb;9(1):4-7. doi: 10.1016/S0952-8180(96)00217-6. PMID 9051538
- [Background] Nunez J, Hughes J, Wareham K, Asai T. Timing of removal of the laryngeal mask airway. Anaesthesia. 1998 Feb;53(2):126-30. doi: 10.1046/j.1365-2044.1998.00298.x. PMID 9534633
- [Background] Pappas AL, Sukhani R, Lurie J, Pawlowski J, Sawicki K, Corsino A. Severity of airway hyperreactivity associated with laryngeal mask airway removal: correlation with volatile anesthetic choice and depth of anesthesia. J Clin Anesth. 2001 Nov;13(7):498-503. doi: 10.1016/s0952-8180(01)00318-x. PMID 11704447
- [Background] Baird MB, Mayor AH, Goodwin AP. Removal of the laryngeal mask airway: factors affecting the incidence of post-operative adverse respiratory events in 300 patients. Eur J Anaesthesiol. 1999 Apr;16(4):251-6. doi: 10.1046/j.1365-2346.1999.00476.x. PMID 10234495
- [Background] Kitching AJ, Walpole AR, Blogg CE. Removal of the laryngeal mask airway in children: anaesthetized compared with awake. Br J Anaesth. 1996 Jun;76(6):874-6. doi: 10.1093/bja/76.6.874. PMID 8679367
- [Background] Afshan G, Chohan U, Qamar-Ul-Hoda M, Kamal RS. Is there a role of a small dose of propofol in the treatment of laryngeal spasm? Paediatr Anaesth. 2002 Sep;12(7):625-8. doi: 10.1046/j.1460-9592.2002.00937.x. PMID 12358660